CLINICAL TRIAL: NCT03530618
Title: Central Line Insertion Technique in Small Infants Using Flexible Tip Straight Guidewire and J-tip Guidewire: a Randomized Controlled Trials
Brief Title: Central Line Catheterization With Flexible Tip Straight Guidewire in Small Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-1803-150-935
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Catheterization, Central Venous

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flexible tip straight guidewire (Experimental)
  Interventions: Device: Flexible tip straight guidewire
- J-tip guidewire (Experimental)
  Interventions: Device: J-tip

INTERVENTIONS:
Device: Flexible tip straight guidewire — Use a flexible tip straight guidewire for ultrasound-guided central venous catheterization
  Arms: Flexible tip straight guidewire
Device: J-tip — Use a J tip straight guidewire for ultrasound-guided central venous catheterization
  Arms: J-tip guidewire

SUMMARY:
The purpose of this study is to compare the differences in central venous catheter insertion time, success rate, and complication between the flexible tip straight guidewire and J-tip guidewire for ultrasound-guided central venous catheterization in small children.

ELIGIBILITY:
Inclusion Criteria:

* surgery under general anesthesia
* require central venous catheterization

Exclusion Criteria:

* central vein anomaly
* hematoma in central vein
* catheterization site infection

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
First successful central venous catheterization rate | Interval between skin penetration of the needle and installation of the indwelling catheter, an expected average of 3 minutes

SECONDARY OUTCOMES:
Time to first puncture of central vein | Interval between skin penetration of the needle and flashback of blood, an expected average of 30 seconds
Time to guide wire insertion | Interval between skin penetration and removal of the needle after guide wire insertion, an expected average of 90 seconds
Total time to central venous catheterization | Interval between skin penetration of the needle and installation of the indwelling catheter, an expected average of 3 minutes
Number of central vein puncture trial | up to 5 times, an expected average observation time of 30 seconds
Number of guide wire insertion trial | up to 5 times, an expected average observation time of 90 seconds
First successful central vein puncture rate | Interval between skin penetration of the needle or angiocatheter and flashback of blood, an expected average of 30 seconds
First successful guide wire insertion rate | Interval between skin penetration and removal of the needle after guide wire insertion, an expected average of 90 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, Professor, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim EH, Kang P, Song IS, Ji SH, Jang YE, Lee JH, Kim HS, Kim JT. Straight-tip guidewire versus J-tip guidewire for central venous catheterisation in neonates and small infants: A randomised controlled trial. Eur J Anaesthesiol. 2022 Aug 1;39(8):656-661. doi: 10.1097/EJA.0000000000001695. Epub 2022 Jul 7. PMID 35793466